CLINICAL TRIAL: NCT06487000
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multi-Center Phase 2 Clinical Trial to Evaluate Efficacy and Safety of EC-18 in Moderate to Severe Atopic Dermatitis
Brief Title: Determine the Dose-dependent Efficacy and Safety of EC-18 in Patients With Moderate to Severe Atopic Dermatitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Enzychem Lifesciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EC-18-205
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EC-18 1000mg (Experimental): [EC-18 2 capsules / Placebo 2 capsules]
  Interventions: Drug: EC-18; Drug: Placebo EC-18
- EC-18 2000mg (Experimental): [EC-18 4 capsules]
  Interventions: Drug: EC-18
- Placebo (Placebo Comparator): [Placebo 4 capsules]
  Interventions: Drug: Placebo EC-18

INTERVENTIONS:
Drug: EC-18 — oral administration, QD
  Other Names: EC-18 soft capsules
  Arms: EC-18 1000mg; EC-18 2000mg
Drug: Placebo EC-18 — oral administration, QD
  Arms: EC-18 1000mg; Placebo

SUMMARY:
To evaluate the efficacy and safety of oral administration of dose-dependent EC-18 for 16 weeks in patients with moderate to severe atopic dermatitis

DETAILED DESCRIPTION:
This study will utilize a randomized, double blind, placebo-controlled, parallel-group, multi-Center design. The Experimental group 1 will receive 1000mg of EC-18[2 capsules of EC-18 500mg, 2 capsules of placebo]. The experimental group 2 will receive 2000mg of EC-18 [4 capsules of EC-18]. The placebo group will receive 4 capsules of placebo. The time frame of this clinical trial will consist 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

At the time of screening:

* aged 19 to under 80 at the time of written consent.
* Patients diagnosed with atopic dermatitis according to the Hanifin and Rajka criteria (≥3 major symptoms out of 4 and ≥3 minor symptoms out of 23) for at least 12 months prior to screening
* Patients requiring systemic therapy for disease control due to either a documented inadequate response to topical drug treatment for at least 4 weeks (within 6 months prior to screening visit), or where topical therapy is medically not recommended (due to significant side effects or safety concerns)
* Patients with Moderate to Severe Atopic dermatitis

  * BSA ≥ 10%
  * EASI score ≥16
  * IGA score ≥3
  * Pruritus NRS score ≥3
* Patients who have been fully informed about this clinical trial, have voluntarily decided to participate, and have provided written consent to faithfully comply with the trial requirements.

At the time of baseline visit

* Signed informed consent
* Patients who have used emollients continuously for the 7 days prior to baseline visit

Exclusion Criteria:

* Patients with serious skin conditions other than atopic dermatitis (e.g. psoriasis, discoid lupus erythematosus, or erythema multiforme that, as judged by the investigator, would adversely affect the evaluation of atopic dermatitis)
* Patients with a history of chronic immunosuppression
* Patients with ongoing malignant tumors at screening or diagnosed within the last 5 years
* Patients who have undergone bone marrow or organ transplantation
* Patients with hypertension (e.g. systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg)
* Patients with ulcerative or erosive lesions
* Patients with Netherton's Syndrome
* Patients with clinically significant severe infections (e.g. infections requiring prolonged antibiotic or immunotherapy treatment) or severe trauma as judged by the investigator
* Patients with positive serum test results at screening (HBs Ag, HCV Ab, HIV Ab). However, patients with a positive HCV Ab result may be eligible if they have achieved HCV RNA negativity after treatment
* Patients at screening (Visit 1) with laboratory test results falling under the following criteria:

  * HbA1c ≥ 7%(Despite medication treatment)
  * ALT and AST ≥ 5 times the upper limit of normal (ULN)
  * eGFR (CKD-EPI_ < 30 ml/ min/1.73m²
  * Serum potassium > 5.5 mEq/L
  * LDL-C >190mg/dL or TC > 500mg/dl (Despite medication treatment)
* Patients with hypersensitivity reactions to the components of the investigational durg or its formulations
* Treatment with topical corticosteroids, local calcineurin inhibitors, topical Janus kinase inhibitors, Tars, antibiotic cream, topical or oral antihistamines within the past 7 days prior to baseline
* Patients who have undergone sunbathing, tanning bed use, ultraviolet B (UVB) therapy, or PUVA (psoralen + ultraviolet A (UVA)) therapy for relief of atopic dermatitis symptoms within the 14 days prior to baseline
* Treatment with systemic immunosuppressants/immunomodulators and/or systemic corticosteroids within the 28 days prior to baseline (patients who have used stable doses of inhaled corticosteroids or nasal sprays for more than 3 months are eligible to participate)
* Patients who have received treatment with biologics other than dupilumab within 3 months prior to baseline.
* Patients who have received treatment with dupilumab within 3 months prior to baseline
* Patients with a history of drug or alcohol abuse within 1 year prior to screening
* Pregnant or breastfeeding women.
* Women who test positive for pregnancy at screening or who plan to become pregnant during the clinical trial period and up to one month after the end of the investigational drug administration, or who do not agree to use appropriate contraception*, and men.

  * Appropriate contraception: complete abstinence, hormonal contraceptives without known drug interactions [levonorgestrel intrauterine system (IUS) (Mirena), medroxyprogesterone], surgical sterilization (vasectomy, bilateral tubal ligation, etc.). Note that periodic abstinence (e.g., ovulation timing, symptothermal method, or post- ovulation) or withdrawal is not considered appropriate contraception.
* Patients who have received any investigational drug within 6 months prior to screening (those who have not received an investigational drug or who have participated in non-interventional observational studies are eligible)
* Other patients deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in EASI score at 16 weeks compared to baseline | Baseline, week 16
  Eczema Area Severity Index (EASI) score: Sum of the 4 region scores (Head/neck, Trunk , Upper extremities, Lower extremities)
  Score range: [0=none ~ 72=very severe]

SECONDARY OUTCOMES:
Change in EASI score at 4, 8, and 12 weeks compared to baseline. | Baseline, week 4, 8, 12
  Eczema Area Severity Index (EASI) score: Sum of the 4 region scores (Head/neck, Trunk , Upper extremities, Lower extremities)
  Score range: [0=none ~ 72=very severe]
Percentage change in EASI score at 4, 8, 12, and 16 weeks compared to baseline | Baseline, week 4, 8, 12, 16
  Eczema Area Severity Index (EASI) score: Sum of the 4 region scores (Head/neck, Trunk , Upper extremities, Lower extremities)
  Score range: [0=none ~ 72=very severe]
Proportion of subjects achieving EASI-50, EASI-75, and EASI-90 at 4, 8, 12, and 16 weeks compared to baseline. | Baseline, week 4, 8, 12, 16
  Eczema Area Severity Index (EASI) score: Sum of the 4 region scores (Head/neck, Trunk , Upper extremities, Lower extremities)
  Score range: [0=none ~ 72=very severe]
Change in IGA score at 4, 8, 12, and 16 weeks compared to baseline. | Baseline, week 4, 8, 12, 16
  Investigator's Global Assessment(IGA) score: [0 = Clear, 1 = Almost clear, 2 = Mild, 3 = Moderate, 4 = Severe]
Proportion of subjects with an IGA score of 0 or 1 and at least a 2-point reduction in IGA score at 4, 8, 12, and 16 weeks compared to baseline. | Baseline, week 4, 8, 12, 16
  Investigator's Global Assessment(IGA) score: [0 = Clear, 1 = Almost clear, 2 = Mild, 3 = Moderate, 4 = Severe]
Change in pruritus NRS score at 4, 8, 12, and 16 weeks compared to baseline. Change in pruritus NRS score at 4, 8, 12, and 16 weeks compared to baseline. Change in pruritus NRS score at 4, 8, 12, and 16 weeks compared to baseline. | Baseline, week 4, 8, 12, 16
  Pruritus Numerical Rating Scale(NRS): The scale of perceived itchiness from [0=none to 10=very severe]
Percentage change in pruritus NRS score at 4, 8, 12, and 16 weeks compared to baseline. | Baseline, week 4, 8, 12, 16
  Pruritus Numerical Rating Scale(NRS): The scale of perceived itchiness from [0=none to 10=very severe]
Proportion of subjects with a pruritus NRS score reduction of 4 points or more at 4, 8, 12, and 16 weeks compared to baseline. | Baseline, week 4, 8, 12, 16
  Pruritus Numerical Rating Scale(NRS): The scale of perceived itchiness from [0=none to 10=very severe]
Change in sleep disturbance NRS score at 4, 8, 12, and 16 weeks compared to baseline. | Baseline, week 4, 8, 12, 16
  Sleep Disturbance Numerical Rating Scale(NRS): The scale of perceived sleep disturbance from [0=none to 10=very severe]
Frequency and duration of application of the rescue medication (tacrolimus ointment). | week 4 ~ week 16

OTHER OUTCOMES:
(Exploratory) Change in DLQI score at 4, 8, 12, and 16 weeks compared to baseline. | Baseline, week 4, 8, 12, 16
  Dermatology Life Quality Index (DLQI) score [0-1] = No effect on patient's life [2-5] = Minimal effect on patient's life [6-10] = Moderate effect on patient's life [11-20] = Very large effect [21 - 30] = Extremely large effect
(Exploratory) Changes in inflammatory biomarker (cytokine) levels at 4, 8, 12, and 16 weeks compared to baseline. | Baseline, weeks 4, 8, 12, 16
  [IL-4, IL-13, IL-6, IFN- γ, IL-17A, IgE]